CLINICAL TRIAL: NCT00719355
Title: Polestriding Versus Walking for PAD Rehabilitation
Brief Title: Polestriding Versus Walking for Subjects With Poor Leg Circulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Eileen G. Collins, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-0477; R01NR008877 (NIH)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Walking; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking with Poles (Experimental): Patients were assigned to a 24 week walking with poles program of rehabilitation. The intervention was the additional of poles to the walking program.
  Interventions: Behavioral: Walking with poles
- Traditional walking program (Active Comparator): Patients were assigned to a 24 week traditional walking program.
  Interventions: Behavioral: Walking exercise

INTERVENTIONS:
Behavioral: Walking with poles — Patients walked with poles, 20-45 minutes, 3 times/week for 24 weeks.
  Other Names: Exercise
  Arms: Walking with Poles
Behavioral: Walking exercise — Patients walked for 20-45 minutes, 3 times/week for 24 weeks.
  Other Names: Exercise
  Arms: Traditional walking program

SUMMARY:
The purpose of this study is to compare the effects of polestriding (walking with poles) and traditional walking on physical endurance in subjects with poor circulation in their legs. Another goal is to evaluate the effectiveness of a walking program in increasing the amount of oxygen in the calf muscles and therefore improving overall physical activity and quality of life.

DETAILED DESCRIPTION:
Peripheral Arterial Disease (PAD/PVD) is caused by decreased blood flow to the legs. The most common symptom is intermittent claudication pain during walking that is relieved by rest. Walking is the primary treatment prescribed for PAD rehabilitation. Polestriding uses muscles of the upper and lower body in a continuous movement. Walking with poles increases stride length, cadence and walking speed and decreases ground reaction forces on the joints. Subjects in this study will participate in a walking program with or without poles.

Dr. Collins' research focuses on physical activity interventions to improve the functional status of persons with chronic illness. Several rehabilitation studies have tested the efficacy of walking exercise for patients with PAD. Studies on polestriding indicate that it may be superior to traditional walking, but these two methods have never been compared. Approximately 30% of patients with coronary artery disease have PAD as their only symptom. As the population ages and more people are affected by this debilitating condition, nurse-initiated rehabilitative therapies, such as polestriding, need to be explored. The consent form explains the purpose of the study in addition to the procedures, risks, benefits, options, confidentiality, costs, and compensation. Participants are also asked to sign a HIPPA authorization.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Vascular Disease
* Cramping/Claudication Pain in legs while walking
* Ankle Brachial Index (measure of circulation by doppler) .90 or less

Exclusion Criteria:

* Ulcers or sores on feet or legs
* Unable to walk or confined to a wheelchair
* Amputations or severe arthritis pain in shoulders, knees, or hips
* Medical conditions which would exclude subject from participating in an exercise program
* Vascular Surgery within the last six months, or planning vascular surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Collins, RN, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Background] Collins EG, Langbein WE, Orebaugh C, Bammert C, Hanson K, Reda D, Edwards LC, Littooy FN. Cardiovascular training effect associated with polestriding exercise in patients with peripheral arterial disease. J Cardiovasc Nurs. 2005 May-Jun;20(3):177-85. doi: 10.1097/00005082-200505000-00009. PMID 15870588
- [Background] Collins EG, Edwin Langbein W, Orebaugh C, Bammert C, Hanson K, Reda D, Edwards LC, Littooy FN. PoleStriding exercise and vitamin E for management of peripheral vascular disease. Med Sci Sports Exerc. 2003 Mar;35(3):384-93. doi: 10.1249/01.MSS.0000053658.82687.FF. PMID 12618567
- [Background] Langbein WE, Collins EG, Orebaugh C, Maloney C, Williams KJ, Littooy FN, Edwards LC. Increasing exercise tolerance of persons limited by claudication pain using polestriding. J Vasc Surg. 2002 May;35(5):887-93. doi: 10.1067/mva.2002.123756. PMID 12021703
- [Result] Fritschi C, Collins EG, O'Connell S, McBurney C, Butler J, Edwards L. The effects of smoking status on walking ability and health-related quality of life in patients with peripheral arterial disease. J Cardiovasc Nurs. 2013 Jul-Aug;28(4):380-6. doi: 10.1097/JCN.0b013e31824af587. PMID 22495802
- [Result] Collins EG, McBurney C, Butler J, Jelinek C, O'Connell S, Fritschi C, Reda D. The Effects of Walking or Walking-with-Poles Training on Tissue Oxygenation in Patients with Peripheral Arterial Disease. Int J Vasc Med. 2012;2012:985025. doi: 10.1155/2012/985025. Epub 2012 Sep 25. PMID 23050152
- [Result] Collins EG, O'connell S, McBurney C, Jelinek C, Butler J, Reda D, Gerber BS, Hurt C, Grabiner M. Comparison of walking with poles and traditional walking for peripheral arterial disease rehabilitation. J Cardiopulm Rehabil Prev. 2012 Jul-Aug;32(4):210-8. doi: 10.1097/HCR.0b013e31825828f4. PMID 22595894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at University of Illinois at Chicago, the Edward Hines Jr., VA Hospital, through radio and print advertising. 146 patients were enrolled in the study and 103 were randomized.
Pre-assignment Details: Patients were screened prior to randomization. Patients were disqualified from the study due to coronary arterial disease, they changed their mind, other medical reasons or it was found that they did not have periphaeral arterial disease.
Groups:
- Walking With Poles: Patients exercised using walking poles, 3 times weekly for 24 weeks.
- Traditional Walking Group: Patients exercised for 24 weeks as part of a traditional walking training group.
Period: Overall Study
Arm/Group | Walking With Poles | Traditional Walking Group
Started | 51 | 52
Completed 6 Weeks | 49 | 48
Completed 12 Weeks | 43 | 46
Completed 24 Weeks | 34 | 43
Completed 32 Weeks | 33 | 39
Completed | 33 | 39
Not Completed | 18 | 13
Not completed — Death | 0 | 1
Not completed — Medical | 14 | 5
Not completed — Compliance | 4 | 6
Not completed — Moved | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking With Poles | Traditional Walking Group | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 22 | 39
  >=65 years | 34 | 30 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 71.4 (9.1) | 68.0 (8.5) | 69.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 47 | 49 | 96
Region of Enrollment [Number; unit: participants]
  United States | 51 | 52 | 103

OUTCOME MEASURES:

1. Primary Outcome: Length of Exercise Duration on the Treadmill Constant Work Rate Exercise Test
Description: Patients walked on the CWR test at 85% of his/her peak VO2 on the baseline progressive treadmill test. Since the polewalking group was older than the walking group, subject age was entered into the analysis as a co-variate. Intent-to-treat (ITT) analyses were used. The last measurement taken for all subjects with at least one follow-up test was carried forward (n=97).
Time Frame: Baseline and 24 weeks
Population: Data were analyzed on patients with at least 1 follow-up treadmill test from baseline.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Walking With Poles | Traditional Walking Group
Number analyzed (Participants) | 49 | 48
minutes | 15.15 (12.31) | 21.40 (16.46)
Statistical Analysis 1: Comparison: Walking With Poles vs Traditional Walking Group; Observed power for our primary analysis was 0.64; Test type: Superiority or Other; p = 0.033, ANCOVA — A priori level of significance was set at p <0.05; Repeated-measures ANCOVA using intent-to-treat procedures, was used for the primary outcome variable. Analyses were adjusted for age; Mean Difference (Final Values) = 6.25, Standard Deviation 14.4

2. Secondary Outcome: Onset of Claudication Pain During Constant Work Rate Treadmill Test
Description: Perceived pain onset was recorded during the constant workrate test using the Borg ratio scale. Patient rated their pain from 0-10. Time elapased on the treadmill (minutes) at the onset of pain was recorded.
Time Frame: At 24 weeks
Population: Data were analyzed on all patients with at least 1 follow up constant workrate treadmill test.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Walking With Poles | Traditional Walking Group
Number analyzed (Participants) | 49 | 48
minutes | 9.3 (12.1) | 6.8 (4.8)
Statistical Analysis 1: Comparison: Walking With Poles vs Traditional Walking Group; Test type: Superiority or Other; p = 0.109, ANCOVA; Repeated measures ANCOVA was used with intent to treat analysis. The co-variant was age; Mean Difference (Final Values) = 1.4, Standard Deviation 3.65

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 32 weeks (the duration of the study).
Arm/Group | Walking With Poles | Traditional Walking Group
Serious Adverse Events (participants affected / at risk) | 4/51 | 6/52
Other Adverse Events (participants affected / at risk) | 2/52 | 3/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Walking With Poles (N=51) | Traditional Walking Group (N=52)
Death (Vascular disorders) | 0 (0) | 1 (1)
Hospitalization respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Includes hospitalizations for pnemonia and upper respiratory tract infections.
Hospitalization renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) — Patient hospitalized for acute renal failure.
Hospitalization cardiac related (Cardiac disorders) | 3 (3) | 1 (1)
Hospitalization bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization low blood sugar (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Walking With Poles (N=52) | Traditional Walking Group (N=51)
Fall (Social circumstances) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to the small number of women in the trial, results cannot be generalized to women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes